CLINICAL TRIAL: NCT00678847
Title: Chronic Venous ULcer TReatment Analyzing Bio-Electrical Stimulation Therapy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kingfisher Healthcare (Industry)
Responsible Party: Dr. Henk Snyman, Kingfisher Healthcare
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ULTRA-BEST
Record Dates: First submitted 2008-03-14; First posted 2008-05-16 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-03

CONDITIONS: Chronic Venous Leg Ulcers
Keywords: bio-electrical stimulation therapy; chronic venous ulcers; microcurrent; chronic wounds; complete healing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Placebo Comparator)
  Interventions: Device: KFH NOVO (inactive) + SCT
- A (Active Comparator)
  Interventions: Device: KFH Novo (BEST) + SCT

INTERVENTIONS:
Device: KFH NOVO (inactive) + SCT — inactive device (placebo) 2 x 1hour/day for total period of 8 weeks + standardized conventional therapy (SCT)
  Other Names: KFH NOVO
  Arms: B
Device: KFH Novo (BEST) + SCT — 2 x 1 hour/day bio-electrical stimulation (BEST) for total period for total period of 8 weeks in combination with standardized conventional therapy (SCT)
  Other Names: KFH Novo
  Arms: A

SUMMARY:
Indication: Subjects with chronic venous leg ulcers

Primary Objective:

• To evaluate the efficacy of bio-electrical stimulation therapy in the healing of chronic venous leg ulcers

Secondary Objective(s):

* To evaluate the percentage of wound healing every two weeks
* To evaluate the complete ulcer healing every two weeks
* To evaluate the time to complete ulcer healing
* To evaluate the recurrence rate at the end of the follow-up period
* To evaluate pain
* To evaluate the quality of life

Study Design and Treatment Scheme:

This is a Kingfisher Healthcare NV sponsored, national, multicenter, randomized, prospective study in which data will be collected of subjects with chronic venous leg ulcers receiving standardized conventional therapy (SCT). Subjects will be randomized into two groups receiving SCT + placebo or SCT + bio-electrical stimulation therapy (BEST) to evaluate the effect of BEST on the wound healing process.

Patients answering the eligibility criteria will receive standardized conventional therapy during 4 weeks before actual study start and will then again be evaluated on eligibility according to wound healing rate. Only patients with a wound surface that has not significantly changed (both increased or decreased) will be randomized in the treatment period.

During the treatment period patients will receive SCT with placebo or SCT in combination with bio-electrical stimulation therapy on a daily basis for two hours, during 8 weeks.

Patients will be in follow-up period for a maximum of 8 weeks after treatment period.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥ 18 years old, male or female
* Before any subject data is collected, the appropriate written informed consent must be obtained (see appendix H).
* Confirmation of venous insufficiency during the last 5 years by Duplex examination
* Chronic venous leg ulcers (>12 weeks) not healing with conventional therapy
* Study ulcer size between 8 to 20 cm² and without clinical signs of infection
* No presence of other ulcers in a radius of 5 cm around the study ulcer
* No surgery for venous insufficiency within the last 6 months
* No arterial insufficiency (ABI between 0,7 and 1,3)
* BMI < 40
* No uncontrolled diabetes or any uncontrolled systemic condition that might impair wound healing
* No decubitus wounds
* Ambulant subject
* Written informed consent

Exclusion Criteria:

* Subjects with implanted electrical devices (e.g. cardiac pacemakers)
* Subjects having a concurrent malignancy or being less than 3 years after the end of their cancer therapy
* Subjects with active osteomyelitis
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of bio-electrical stimulation therapy in the healing of chronic venous leg ulcers | every two weeks during treatment (8 weeks) and twice during follow-up period (8 weeks)

SECONDARY OUTCOMES:
To evaluate pain | every two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mieke Flour, MD, Study Chair — UZ Gasthuisberg, Leuven (Belgium); Michel de la Brassinne, MD, Principal Investigator — CHU Sart Tilman, Liege (Belgium); Bert Boyden, MD, Principal Investigator — Virga Jesse Ziekenhuis, Hasselt (Belgium); Hilde Beele, MD, Principal Investigator — UZ Gent, Belgium; Diane Roseeuw, MD, Principal Investigator — UZ Brussel (Belgium)
Locations (1):
- UZ Gasthuisberg, Leuven, Belgium